CLINICAL TRIAL: NCT00117429
Title: A Phase I, Randomized, Double-Blind Clinical Trial of the HIV gp120/NefTat/AS02A Vaccine Candidate in Subjects With Well-Controlled Chronic HIV-1 Infection on Highly Active Antiretroviral Therapy (HAART)
Brief Title: Study of the HIV gp120/NefTat/AS02A Vaccine to Treat Individuals With Chronic HIV-1 Infection on Highly Active Antiretroviral Therapy (HAART)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Marcus Altfeld, M.D., Ph.D. (Individual)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Marcus Altfeld, Massachusetts General Hosptial
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PARC001; GSK: TH-HIV-007
Record Dates: First submitted 2005-06-30; First posted 2005-07-07 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-02

CONDITIONS: HIV Infections
Keywords: HIV-1; therapeutic vaccination; cellular immunity; humoral immunity; HAART; chronic HIV-1 infection; Treatment Experienced; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections | interventions — HIV Envelope Protein gp120

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Biological: HIV gp120/NefTat/AS02A Vaccine — im injection, 0.6-0.7 ml

SUMMARY:
This study will test the safety and immunogenicity of the gp120/NefTat/AS02A vaccine candidate in individuals with chronic HIV-1 infection successfully treated with HAART. The rationale for this study is based on previous scientific experiments, including data indicating that this vaccine can elicit strong HIV-1-specific T cell immune responses in humans and monkeys and lead to a retardation of HIV-1 disease progression in animal models of HIV-1 infection.

The HIV vaccine to be administered during this study consists of three recombinant HIV clade B viral antigens: the envelope glycoprotein gp120 and two regulatory proteins, Nef and Tat.The antigens are formulated in a proprietary adjuvant, AS02A, comprised of two immunostimulants in an oil-in-water emulsion (gp120/NefTat/AS02A). The vaccine and the adjuvant are manufactured and provided for the study by GlaxoSmithKline Biologicals, Rixensart, Belgium. The drugs will be given by intramuscular (IM) injection at a standard dose of 20 mg together with 0.5 ml of the AS02A adjuvant.

Twenty HIV-1 infected individuals will be randomly enrolled into three different study groups, receiving either the gp120/NefTat/AS02A vaccine (10 individuals), the AS02A adjuvant alone (5 individuals) or a placebo (5 individuals). After obtaining informed consent, subjects will have a history and physical exam performed and have laboratory tests to confirm they meet all inclusion and exclusion entry criteria. Women of childbearing potential will have a pregnancy test prior to each injection of the investigational product. Injections with vaccine, adjuvant alone, or placebo will then be performed at weeks 0, 4, and 12. Study participants will undergo close monitoring after each vaccination. Blood samples will be obtained for immunological assays at study baseline (2 times) and weeks 2, 4, 6, 12, 14, 24, and 48. All patients will maintain their antiretroviral treatment regimen during the entire study period.

DETAILED DESCRIPTION:
DESIGN: This study is a randomized, double blind clinical trial of the gp120/NefTat/AS02A vaccine in individuals with well-controlled chronic HIV-1 infection who have been successfully treated with highly active antiretroviral therapy (HAART). The adjuvanted protein vaccine candidate consists of three recombinant viral antigens: the envelope glycoprotein gp120 and two regulatory proteins, Nef and Tat. The latter are expressed as one recombinant fusion protein, NefTat. The antigens are formulated in the proprietary AS02A adjuvant. The goal of this trial is to assess the safety and immunogenicity of the gp120/NefTat/AS02A vaccine in HIV-1-infected individuals.

DURATION: 48 weeks

SAMPLE SIZE: 20 subjects

POPULATION: Subjects with chronic HIV-1 infection receiving highly active antiretroviral therapy (HAART) with HIV RNA levels <50 copies/mL on at least two measurements in the previous 6 months and a CD4+ T cell count >400 cells/mm3 within 45 days of study entry will be eligible for this study.

REGIMEN: Enrolled patients will be randomized to receive either the vaccine (gp120/NefTat/AS02A) (10 individuals), the AS02A adjuvant only (5 individuals) or a placebo (5 individuals). Injections will be administered IM at weeks 0, 4, and 12.

OBJECTIVES: The two primary objectives of this study are:

* to evaluate the safety and tolerability of the gp120/NefTat/AS02A vaccine in individuals with well-controlled chronic HIV-1 infection on HAART; and
* to evaluate the cell-mediated immune response (IL-2 secreting CD4+ T cells) to at least one vaccinal antigen induced by the vaccine-adjuvant combination in individuals with chronic HIV-1 infection on successful HAART, at two weeks after the third vaccination.

ENDPOINTS: The two co-primary study endpoints will be:

* the occurrence, intensity, and relationship of any local and general signs and symptoms during a 7-day follow-up period after each vaccination (primary safety endpoint); and
* the changes in the frequency of IL-2 secreting CD4+ T cells in response to at least one vaccinal antigen (primary immunogenicity endpoint) in the three different patient categories, assessed two weeks after the third vaccination.

ELIGIBILITY:
Inclusion Criteria:

The study will include subjects who meet all of the following criteria:

* Male or female, between 18 to 60 years of age at the time of the first vaccination
* Informed consent signed prior to all study procedures
* No evidence of acute HIV seroconversion in the 12 months prior to the initiation of antiretroviral therapy
* Receiving a potent antiretroviral drug regimen for a minimum of 12 consecutive months prior to screening with no interruption of therapy for > 2 weeks.

A potent antiretroviral drug regimen is defined as any of the following: *two nucleoside reverse transcriptase inhibitors with either a protease inhibitor or a non-nucleoside reverse transcriptase inhibitor; *a boosted protease inhibitor with either one or two nucleoside reverse transcriptase inhibitors or a non-nucleoside reverse transcriptase inhibitor.

* Documented suppressed HIV-1 RNA. Subjects must have plasma HIV-1 RNA values <50 copies/ml on at least two measurements during the 6 months prior to the study entry.
* CD4+ T cell count >400 cells/mm3 within 45 days of the first vaccination
* CD4 count >200 cells/mm3 at all times
* Laboratory values within 45 days prior to the first vaccination that meet the following criteria:

  * Hemoglobin >9.0 g/dL;
  * Absolute neutrophil count ≥ 1000/mm3;
  * Platelet count ≥ 75,000/mm3;
  * Prothrombin time (PT) < 1.2 x upper limit of normal (ULN) and partial thromboplastin time (PTT) < 1.5 x ULN;
  * Total serum creatinine < 1.3 x ULN;
  * Total serum bilirubin < 2.0 x ULN;
  * Alkaline phosphatase, AST (SGOT) and ALT (SGPT) < 1.5 x ULN.
* Negative serologic test for HBsAg
* Negative serologic test for antibodies to HCV or negative HCV PCR if anti-HCV antibodies are positive.
* Female patient of childbearing potential must:

  * Have a negative urine pregnancy test (sensitive to 25 IU HCG) immediately prior to vaccination;
  * Have no intention of conceiving during the entire study period;
  * Agree to use an effective method of birth control during the entire study period. Effective methods of birth control include:

    1. Condoms (male or female) with or without spermicidal agent. Condoms are recommended because their appropriate use is the only contraception method effective for preventing HIV transmission;
    2. Diaphragm or cervical cap with spermicide;
    3. Intrauterine device (IUD). An IUD is an adequate method of birth control, but increases the risk of pelvic inflammatory disease;
    4. An FDA-approved oral contraceptive, provided there is no interaction with the woman's current antiretroviral therapy or other medications;
  * If participating in sexual activity that could lead to pregnancy, the male subject or his partner must also use contraception.

Exclusion Criteria:

* HIV-1 RNA > 50 copies/mL within 6 months of screening.
* Received antiretroviral therapy within 12 months of known HIV-1 seroconversion.
* History of clinically significant cardiac, pulmonary, gastrointestinal, hepatic, renal, pancreatic, or neurological disease
* Recent (<24 hours) febrile illness on the day of vaccination (temperature >101 degrees F, oral)
* History of CD4 count <200 cells/mm3.
* Female subject who is pregnant or nursing a child
* Received any immune globulin or blood products within 3 months prior to vaccination or plans to receive such products during the study
* Received any live vaccine within 30 days prior to study vaccination or any inactivated vaccine within 14 days prior to study vaccination
* Previously participated in any HIV vaccine clinical trial (unless it is documented that the subject received only placebo)
* History of any AIDS defining illness
* Any change in antiretroviral drug regimen within 12 weeks prior to screening
* Use of any immunomodulatory agents within 30 days prior to study enrollment or planned use during the trial
* Active drug or alcohol use or dependence that, in the opinion of the sponsor, would interfere with adherence to study requirements.
* Any condition or history of illness which, in the opinion of the investigator, might interfere with the evaluation of the study objectives
* Subject has a history of anaphylaxis to any vaccine
* Subject has a history of allergy to any adjuvant component
* Subject is taking any of the following medications: systemic steroids (inhaled or nasal steroid therapy is permitted), interleukins, systemic interferons (e.g. local injection of interferon alpha for treatment of HPV is permitted) or systemic chemotherapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-06; Primary Completion 2007-09 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Occurrence, intensity and relationship of any local and general signs and symptoms during a 7-day follow-up period (i.e. day of vaccination and 6 subsequent days) after each vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Altfeld, MD/PhD, Principal Investigator — Massachusetts General Hospital; Mathias Lichterfeld, MD/PhD, Principal Investigator — Massachusetts Genral Hosptial
Locations (1):
- Massacusetts General Hospital -Infectious Disease Unit, Boston, Massachusetts, United States